CLINICAL TRIAL: NCT06849804
Title: Comparing the Efficacy of Ultrasound Guided Erector Spinae Plane Block, Ultrasound Guided Caudal Block, and Local Infiltration for Postoperative Pain Control in Pediatric Patients Undergoing Unilateral Inguinal Hernia Repair as a Day-Case Surgeries: A Randomized Controlled Trial
Acronym: ECLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Zakarea Wfa, Assisted professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 36264PR1045/1/25
Record Dates: First submitted 2025-02-09; First posted 2025-02-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Group E : erector spinae block ultrasound guided Group C: ultrasound guided caudal block Group L: local infiltration
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group E (Active Comparator): Ultrasound guided erector spinae block
  Interventions: Procedure: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®)
- Group C (Active Comparator): Ultrasound guided caudal block
  Interventions: Procedure: Caudal Block Anesthesia
- Group L (Active Comparator): Local infiltration of the wound
  Interventions: Procedure: Local infiltration in the wound

INTERVENTIONS:
Procedure: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) — Group E (n=25): Erector spinae plain block group will receive 0.5 ml/kg of 0.25%bupivacaine.
  Arms: Group E
Procedure: Caudal Block Anesthesia — Caudal block group will receive 1 ml/kg of 0.25% bupivacaine
  Arms: Group C
Procedure: Local infiltration in the wound — Local Infiltration Group will receive 0.2 ml/kg 0.25% bupivacaine
  Arms: Group L

SUMMARY:
The aim of this study is to evaluate the efficacy of ultrasound guided Erector block versus caudal block versus local wound infiltration perioperatively according to:

Primary outcome: to assess and compare the postoperative analgesic effect using pain score:

Faces Legs Activity Cry Consolability tool (FLACC, 0- 10) at 15 min, 30 min and 1, 2, 3 and 4 h after operation

Secondary outcomes:

First dose of fentanyl as a rescue analgesia in dose of 0.5 μg/kg. Total doses of fentanyl as a rescue analgesia. Demographic data: age, sex, weight, ASA class. Hemodynamic parameter (MAP in (mm/hg) and heart rate (beats/minute)) Motor function will be assessed using the following scale: 0, no motor block; 1, able to move legs; 2, unable to move legs.

Assessment of sedation will be done with objective score based on eye opening: 0- spontaneously, 1- on verbal stimulation, 2- on physical stimulation Adverse events: bradycardia, hypotension, respiratory depression, local anesthesia toxicity, subarachnoid injection in caudal block, PONV, agitation, or urinary catheterization.

DETAILED DESCRIPTION:
This randomized double-blinded study will be carried out on 75 pediatric patients of both sexes undergoing elective unilateral inguinal hernia surgeries in Tanta University Hospitals for a period of from December 2024 to March 2025.

Informed written consent will be obtained from the parents. They will receive an explanation of the purpose of the study, and every patient will have a secret code number. All data of the patients will be confidential with secret codes and private file for each patient, all given data will be used for the current medical research only.

Any unexpected risks that appeared during the research will be cleared to the participants and ethical committee on time. Investigator who is blinded to group allocation provided postoperative care and assessments. Postoperative pain will be assessed. Motor functions and sedation will be assessed as well.

Inclusion Criteria: pediatric patients of both sexes undergoing elective unilateral inguinal hernia surgeries aged from 2 year to 7 years belonging to ASA I or II.

Exclusion Criteria:

Parents refusal. Coagulopathy. Allergy to local anesthesia. Local infection at the site of injection. Neurological anomalies.

Randomization and blindness:

Computer-generated randomization numbers will be used for random allocation and each patients' code will be kept in an opaque sealed envelope. Patients will be randomly allocated with 1:1:1 allocation ratio into three groups in a parallel manner:

Group E (n=25): Erector spinae plain block group will receive 0.5 ml/kg of 0.25%bupivacaine.

Group C (n=25): Caudal block group will receive 1 ml/kg of 0.25% bupivacaine. Group L (n=25): Local Infiltration Group will receive 0.2 ml/kg 0.25% bupivacaine

Methods:

Preoperative:

Medical and surgical history of the patients will be taken, clinical examination of the patients will be performed and routine laboratory investigations as CBC, and coagulation studies.

Intraoperative:

Monitoring (non-invasive blood pressure, pulse oximetry, electrocardiogram and temperature probe) will be applied during induction and maintenance of anesthesia. No premedication will be administered. Anesthesia will be induced with of sevoflurane in 100% oxygen. The intravenous line will be inserted, inject propofol 1-2 mg/kg and airway will be established by using a laryngeal mask airway (LMA). Anesthesia will be maintained with sevoflurane, O2 to Air 50%: 50%, hemodynamic will be adjusted accordingly with a goal of 80-120% baseline arterial pressure and 4.7-6 kPa end-tidal carbon dioxide (EtCO2). Spontaneous breathing will be maintained during surgery. After completion of surgery, the LMA will be removed, and the child will be sent to a post-anesthetic care unit (PACU) so long as there will be no compromise in airway or hemodynamic instability perioperatively.

In group E: A unilateral block will be performed in the lateral decubitus position, with the patient turned on his/her side so that the blocked side will be facing up. Using strict sterilization techniques, the skin will be sterilized with povidone-iodine at the site of needle entry. The level of the 10th thoracic vertebrae will be determined on ultrasound. The ultrasound transducer will be placed at the mid-vertebral line in the sagittal plane. The transducer will be shifted 3.5-4 cm laterally from midline to the surgical side to visualize the erector spinae muscle and transverse process. Using the in-plane technique, the needle will be advanced until the transverse process will be reached. The correct location of the needle tip in the fascial plane deep to the erector spinae muscle will be conﬁrmed by injecting 0.5-1 ml of saline and observing the ﬂuid lifting the erector spinae muscle off the transverse process while avoiding muscle distension (hydro dissection). Once the needle will be at the correct location, a negative aspiration test will be confirmed. Bupivacaine 0.25% at a dose of 0.5 ml/kg will be then injected. The distribution of the injectate within the fascial plane will be observed. The patient will be then placed in the supine position, and we will wait 15 min before beginning of surgery.

In group C: After induction of anesthesia, children from Group C for a right-handed provider, place the patient in the left lateral position (hips and knees flexed). Place the patient in the right lateral position if the provider is left-handed. Prepare the field with sterilizing solution(povidone-iodine) and a sterile drape. Cover the ultrasound probe in a sterile cover. Initial scanning in the transverse plane allows for visualization of the midline and identification of the sacrococcygeal ligament between the 2 sacral cornua. The 2 cornua resemble the 2 eyes of a frog and thus are collectively called the frog-eye sign. The probe will be then rotated 90 degrees to acquire a longitudinal view. The needle will be advanced at a 20-degree angle with needle tip and length visualization. A pop can be appreciated as the needle passes through the sacrococcygeal ligament.

Once the needle will be confirmed to be in the caudal space on the screen, carefully aspirate to confirm absence of CSF or blood. The use of a saline bolus (0.1-0.2 mL/kg) can be performed to confirm correct positioning. If this is the case, real-time visualization of cranial spread of the saline with anterior displacement of the posterior dura will be seen. Lack of dural displacement can be associated with intrathecal or intravascular injection requiring repositioning of the needle. A slow injection of the local anesthetic can then be performed. Wait 15 min before beginning of surgery.

In group L: The patients will be received local infiltration of the surgical area with 0, 25% bupivacaine 10 min before skin incision. The infiltration technique will be standardized as follows: the subcutaneous tissue in the proposed area will be infiltrated with 0.25% bupivacaine before incision. A 16-mm 26-gauge needle will be inserted in the center of the area, and the medial and lateral parts of the proposed skin incision will be infiltrated. The needle still in central position, a fan-shaped application will be administered under the external abdominal fascia. We will wait 15 min before beginning of surgery.

Postoperative: Surgery will be initiated ten minutes after performing the erector spinae block, caudal block or local infiltration. Failure of block will be considered if the patient moves his or her limbs, increase heart rate, mean arterial pressure, or both of more than 15% will be compared with baseline during the surgery. In such instances, the patient will be withdrawn from the study and will be treated with 1-2 μg/kg of fentanyl.

Another investigator who will be blinded to group allocation provided postoperative care and assessments. Postoperative pain will be assessed using Faces Legs Activity Cry Consolability tool (FLACC, 0- 10) at 15 min, 30 min and 1, 2, and 3 h after operation. A child with a score of more than 4 on FLACC received 0.5 μg/kg of fentanyl intravenous for rescue analgesia.

Motor function will be assessed using the following scale: 0, no motor block; 1, able to move legs; 2, unable to move legs. Assessment of sedation will be done with objective score based on eye opening: 0- spontaneously, 1- on verbal stimulation, 2- on physical stimulation. The presence of other adverse events will be evaluated as well including bradycardia, hypotension, respiratory depression, local anesthesia toxicity PONV, agitation, or urinary catheterization. Hypotension and respiratory depression are defined as 80% of baseline arterial pressure and ≤ 95% of pulse oxygen saturation, respectively. The decision to place a urinary catheter for urinary retention and the evaluation of micturition will be made by a urologist. Analgesia on ward will be provided with oral acetaminophen (15 mg/kg).

Children will be discharged from the hospital after 4 to 6 h if they will meet the following discharge criteria: conscious, hemodynamically stable, tolerating oral intake, voiding, walking in an appropriate manner for age, with the absence of side-effects.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria: pediatric patients of both sexes undergoing elective unilateral inguinal hernia surgeries aged from 2 year to 7 years belonging to ASA I or II.

Exclusion Criteria:

Parents refusal. Coagulopathy. Allergy to local anesthesia. Local infection at the site of injection. Neurological anomalies.

Exclusion Criteria:

-

Ages: 24 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Faces Legs Activity Cry Consolability tool (FLACC, 0- 10) at 15 min, 30 min and 1, 2, 3 and 4 h after operation | 4 hours

SECONDARY OUTCOMES:
Analgesic effect of the block | 4 hours
  First dose of fentanyl as a rescue analgesia in dose of 0.5 μg/kg. Total doses of fentanyl as a rescue analgesia. Motor function sedation score based on eye opening: 0- spontaneously, 1- on verbal stimulation, 2- on physical stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Zakarea Wfa, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided